CLINICAL TRIAL: NCT02532725
Title: Relationship of Occupational Heat Stress Endurance, Work, and Percentage of Body Fat in Middle Aged Men
Brief Title: Work-Related Effects of Heat, Activity, and Fat in Middle Aged Men
Status: Completed | Type: Observational
Sponsor: Freeman-Sheldon Research Group, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1120-6134
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Gender; Problem of Aging
Keywords: heat stress response; cardiopulmonary exercise test; men; middle aged; heat-shock response
MeSH Terms: conditions — Obesity; Coitus; Multiple Endocrine Neoplasia Type 1 | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lean: Men aged 35-55 years, having <20% body fat
  Interventions: Procedure: Cardiopulmonary Exercise Stress Test; Procedure: Climatic-Controlled Cardiopulmonary Exercise Stress Test; Procedure: Body Composition Evaluation; Procedure: Pre-Exercise Risk Assessment
- Obese: Men aged 35-55 years, having >29% body fat
  Interventions: Procedure: Cardiopulmonary Exercise Stress Test; Procedure: Climatic-Controlled Cardiopulmonary Exercise Stress Test; Procedure: Body Composition Evaluation; Procedure: Pre-Exercise Risk Assessment

INTERVENTIONS:
Procedure: Cardiopulmonary Exercise Stress Test — Test preceded by warm-up treadmill walking 5 min at 4.8 km/h, 5% grade with a 1 min sitting rest period. Test, then, begins at 4.8 km/h, 2.5% grade with incremental grade increases every 2 min until exhaustion. Ambient environment is maintained at neutral, with effective temperature of 19-21° C. Heart, lungs, temperature, and sweating is monitored during testing.
  Other Names: Progressive Exercise Test; Graded Exercise Test; Stress Test
Procedure: Climatic-Controlled Cardiopulmonary Exercise Stress Test — Test includes 30 min walking bouts on the treadmill, with two 5 min sitting rest periods between bouts (Rest I and Rest II) and 15 min sitting recovery period (Rest III), in effective temperatures of 21.1 (baseline), 26.7, 29.4, 32.2, and 35.0° C. Heart, lungs, temperature, and sweating is monitored during testing.
  Other Names: Environmental Chamber Exercise Test
Procedure: Body Composition Evaluation — Multiple methods are used to accurately estimate percentage of body mass (weight) composed of fat, muscle, bone, and other connective tissues. Four different methods, including caliper and hydrostatic (underwater weighing) are used in this study to ensure an accurate estimation.
Procedure: Pre-Exercise Risk Assessment — Includes non-invasive measurements of body functioning, a physical examination by a physician, and blood and urine testing to select subjects who can exercise with relative safety.
  Other Names: Pre-Participation Examination

SUMMARY:
Obesity is associated with many undesirable health effects and disease, and middle age is associated with increased risk for disease. Unfortunately, while others have looked at the effects of obesity, gender, and middle age, the combined effects of obesity and middle age on men's ability to do work in hot industrial environments have not been satisfactorily investigated.

This small study evaluates the heat tolerance of lean and obese middle aged men both while exercising and resting and the ways in which each compensate for and dissipate increasing environmental heat and heat generated by the body while exercising.

As obesity is a worldwide public health crisis and as populations in many industrialized nations age, it is important to understand the combined effects of obesity and middle age for men on their ability to safely work in hot environments. Such information will permit establishing and revising of safe work standards and inform public health outreach to the target population, itself.

DETAILED DESCRIPTION:
The present study was initially approved by and conducted at The Pennsylvania State University in 1972 for the senior author's (Rodger J McCormick) D.Ed. thesis in Biological Sciences; funding support was provided by the US National Institute of Arthritis, Metabolism, and Digestive Diseases Grant AM-08311 and National Institutes of Health Grant 01748. Data re-analysis and representation of that study was first approved in 2011 by and conducted at the FSRG deGruyter-McKusick Institute of Health Sciences for partial fulfillment of an MS in Clinical and Applied Physiology being pursued by the junior author (Mikaela I Poling). No funding was received for this use of existing data.

Importance of Present Study:

Several heat tolerance studies, including Kenny, Gagnon, Dorman, Hardcastle, and Joy (2010), have indicated that middle-age men can perform hard work in hot environments nearly as well as younger men. Dufour and Candas (2007), in comparing passive heat responses and sudomotor function in young, middle aged, and older men, found only local, not global, decreases in sweat gland output in the two older groups, suggesting at least some significant preservation of sudomotor function. Since most studies employed subjects with lean normal body types, their results in terms of physiological reactions to heat stress may not be applicable to obese middle aged men. Other studies have demonstrated degraded heat stress exercise capacity in obese persons.

Within high heat stress areas such as in the steel, fiberglass, aluminium, mining, professional sports, and defense industries, lean and obese middle aged men can readily be observed performing the same work task in the same hot environment. Little attention has been given to differences between the lean and obese middle aged men in their physiological responses to the combination of internal heat production from the work task performed and the heat load imposed from the external environment.

In the present study, occupational heat stress endurance differences between lean and obese middle aged men and effect of obesity are investigated under laboratory simulated conditions to test the following hypotheses: (1) with greater baseline cardiovascular demands, it is expected that obese middle aged men will have reduced environmental heat tolerance and will gain and store more total heat; (2) poorer environmental heat tolerance of obese middle aged men will be greatly magnified by work (producing added metabolic heat); (3) lean middle aged men will thermoregulate well; (4) lean middle aged men will show few, if any, major signs of inability to compensate for added cardiovascular demands; (5) obese middle aged men will be functioning at a higher percentage of their maximal ventilation of expired oxygen; and (6) obese middle aged men will have poorer pulmonary fitness, as measured by maximal ventilation of expired oxygen, than lean middle aged men.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent and to complete minimum study procedures, as defined by the protocol
* Non-invasive resting blood pressure within normal limits
* Resting electrocardiogram within normal limits
* Hematology and Chemistry (blood) panels within normal limits
* Urinalysis (pH, glucose, and protein) within normal limits
* Negative cardiopulmonary stress test
* Absence of acute or chronic metabolic, cardiovascular, pulmonary, and orthopedic disease

Exclusion Criteria:

* Unable or unwilling to give consent or to complete minimum study procedures, as defined by the protocol
* Non-invasive resting blood pressure outside normal limits
* Resting electrocardiogram outside normal limits
* Hematology and Chemistry (blood) panels outside normal limits
* Urinalysis (pH, glucose, and protein) outside normal limits
* Positive cardiopulmonary stress test
* Presence of acute or chronic metabolic, cardiovascular, pulmonary, and orthopedic disease

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lean and obese middle aged men unaccustomed to working in hot industrial conditions
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 1972-06; Primary Completion 1972-12 (Actual); Study Completion 1972-12 (Actual)

PRIMARY OUTCOMES:
Core (Rectal) Temperature Change with Exercise Level and Increased Heat Load | Evaluated during each session at rest and while exercising, with sessions lasting approximately 165-170 min
  Failure to maintain rectal temperature within 0.15° C of subject baseline for interval from end of exercise Bout 2 to Bout 3.
Oxygen Consumption Change with Exercise Level and Increased Heat Load | Evaluated near the end of Exercise Bout 1 (2 min) and 3 (2 min)
  Oxygen consumption, measured by ventilation of expired oxygen, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by obesity.
Heart rate Change with Exercise Level and Increased Heat Load | Evaluated during each session at rest and while exercising, with sessions lasting approximately 165-170 min
  Increased heart rate, measured electrocardiographically, is used as an index of cardiovascular strain imposed by needs during exercise and exaggerated by obesity.
Difference in Routine and Maximal Ventilation of Expired Oxygen at Neutral Ambient Temperature | Cardiopulmonary Stress Test, during the last 1 min of warm-up and at end of progressive portion as volitional exhaustion approached
  Warm-up approximates steady, normal work, while the progressive portion of the text places maximal metabolic burden on the subject in order to measure upper limit of heart and lung function

SECONDARY OUTCOMES:
Perceived Exertion Change with Exercise Level and Increased Heat Load | Evaluated during each session at rest and while exercising, with sessions lasting approximately 165-170 min
  Increased perceived exertion is used as an index of fatigue, an indirect indicator of physiological strain.
Non-Invasive Arterial Blood Pressure Change with Exercise Level and Increased Heat Load | Evaluated at rest before exercise (20-25 min) and at Rest I (5 min), II (5 min), and III (15 min)
  Increased non-invasive arterial blood pressure rate is used as an index of cardiovascular strain imposed by needs during exercise, is an important indicator of possible onset of shock, and exaggerated by obesity.
Heart Rhythm Change with Exercise Level and Increased Heat Load | Evaluated during each session at rest and while exercising, with sessions lasting approximately 165-170 min
  Heart rhythms, monitored by electrocardiograph, are used as an index of cardiovascular strain imposed by needs during exercise and could be exaggerated by obesity.
Metabolic Rate Change with Exercise Level and Increased Heat Load | Evaluated near the end of Exercise Bout 1 (2 min) and Bout 3 (2 min).
  Rate of energy usage of the body calculated from ventilation of expired oxygen values
Heat Load Change with Exercise Level and Increased Environmental Temperature | During Rest I (5 min), II (5 min), and III (15 min)
  Calculated metabolic and environmental heat gain minus heat loss

OTHER OUTCOMES:
Body Composition | Evaluated before exercise (20 min)
  Body composition, measured by calliper, together with direct indices of physiological strain, is used to determined metabolic and heat storage burden
Age at Death or Current Age | up to 526 months
  Total years alive, not survival after study participation

CONTACTS AND LOCATIONS:
Overall Officials: Rodger J McCormick, DEd, Principal Investigator — Freeman-Sheldon Research Group, Inc.
Locations (1):
- Freeman-Sheldon Research Group, Inc. Headquarters, Buckhannon, West Virginia, United States

REFERENCES:
- [Background] Haymes EM, McCormick RJ, Buskirk ER. Heat tolerance of exercising lean and obese prepubertal boys. J Appl Physiol. 1975 Sep;39(3):457-61. doi: 10.1152/jappl.1975.39.3.457. PMID 1176412
- [Background] Kenny GP, Gagnon D, Dorman LE, Hardcastle SG, Jay O. Heat balance and cumulative heat storage during exercise performed in the heat in physically active younger and middle-aged men. Eur J Appl Physiol. 2010 May;109(1):81-92. doi: 10.1007/s00421-009-1266-4. Epub 2009 Nov 3. PMID 19885672
- [Background] Dufour A, Candas V. Ageing and thermal responses during passive heat exposure: sweating and sensory aspects. Eur J Appl Physiol. 2007 May;100(1):19-26. doi: 10.1007/s00421-007-0396-9. Epub 2007 Jan 23. PMID 17242944
- See also: Freeman-Sheldon Research Group, Inc. (Sponsor's general website) — http://fsrgroup.org